CLINICAL TRIAL: NCT05290948
Title: Comparison of Combined Intravitreal Bevacizumab and Oral Acetazolamide Versus Intravitreal Bevacizumab Alone for the Treatment of Macular Edema Secondary to Retinal Vein Occlusions
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Zahra Rabbani Khah, Head of Ophthalmic Research Center, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14003
Record Dates: First submitted 2022-03-12; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — Acetazolamide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- investigate of the effect of intravitreal injection of bevacizumab with acetazolamide tablets (Active Comparator)
  Interventions: Drug: intravitreal injection of bevacizumab with acetazolamide tablets
- Investigate the effect of intravitreal injection of bevacizumab alone (Active Comparator)
  Interventions: Drug: intravitreal injection of bevacizumab

INTERVENTIONS:
Drug: intravitreal injection of bevacizumab with acetazolamide tablets — intravitreal injection of bevacizumab with acetazolamide tablets
  Arms: investigate of the effect of intravitreal injection of bevacizumab with acetazolamide tablets
Drug: intravitreal injection of bevacizumab — intravitreal injection of bevacizumab
  Arms: Investigate the effect of intravitreal injection of bevacizumab alone

SUMMARY:
In this study, which will be performed as a randomized clinical trial, all patients with macular edema with central involvement (central macular thickness greater than 300 μm) and corrected vision less than or equal to 20/40 and better than 20/400 were included in the study. After a thorough eye examination, people are randomly divided into two groups. The first group was treated with intravitreal injection of Bevacizumab in three injections one month apart with receiving oral Acetazolamide tablets of 250 mg twice a day, and the second group was treated with intravitreal injection of Bevacizumab for three Loads are spaced one month apart. Ophthalmologic examinations and corrected visual acuity, as well as macular thickness examination, are repeated with Spectral-domain Optical coherence tomography (SD-OCT) at the beginning of treatment and at the end of the first, second, and third months. At the end of the study, the rate of changes in visual acuity and macular thickness in the eyes in the two groups will be compared and will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* 20 / 400≤ Best Corrected Visual Acuity ≤20 / 40
* Central macular thickness <300 μm
* The onset of the disease is less than three years
* No other eye diseases that affect the evaluation and process of this study.

Exclusion Criteria:

* It is not possible to provide informed consent.
* Patients who are prohibited from taking oral acetazolamide (renal failure, hepatic failure, history of allergies)
* Other eye diseases that affect the evaluation and process of this study. Including diabetes retinopathy
* History of retinal laser photocoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Estimated)
Dates: Start 2022-03-12 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | 3 months
  the best corrective vision correction that achieved by glasses, as measured on the standard Snellen eye chart

SECONDARY OUTCOMES:
Central macular thickness | 3 months
  Thickness measurements by spectral-domain optical coherence tomography systems (SD-OCT)

CONTACTS AND LOCATIONS:
Locations (1):
- Ophthalmic Research center, Tehran, Iran

REFERENCES:
- [Derived] Karimi S, Nikkhah H, Nafisi H, Nouri H, Ansari I, Barkhordari S, Samnejad S, Abtahi SH. Acetazolamide and bevacizumab combination therapy versus bevacizumab monotherapy in macular edema secondary to retinal vein occlusion. J Fr Ophtalmol. 2023 Apr;46(4):322-326. doi: 10.1016/j.jfo.2022.09.025. Epub 2023 Feb 2. PMID 36739258